CLINICAL TRIAL: NCT02390596
Title: A Phase IIa Multicenter Trial to Assess the Efficacy, and Safety of Anakinra in Patients With Intravenous Immunoglobulin-resistant Kawasaki Disease
Brief Title: Anakinra and Kawasaki Disease
Acronym: KAWAKINRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOM13520; 2014-002715-41 (EudraCT Number)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2018-09

CONDITIONS: Kawasaki Disease; Children
Keywords: Kawasaki disease; anti Interleukin 1 treatment; anakinra; resistance to IVIg; coronary aneurysms; phase II trial
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra (Experimental)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — The dose of Anakinra will be 2mg/kg (patients <10kg and/or <8 months: 4mg/kg). If the patient remains febrile (fever >38°C), he will receive a double dose of anakinra 4mg/kg (patients <10kg and/or <8 months: 6mg/kg) at day1 instead of 2mg/kg. If the patient does not respond to the 4mg/kg dose at visit 3; d1 within 24 hours, he will receive at visit 4; d2, 6mg/kg of anakinra (patients <10kg and/or <8 months: 8mg/kg). Treatment will be continued until they have achieved complete response as defined in the outcome measurement section, and during a maximum of 15 days.
  Other Names: Kineret

SUMMARY:
The study is designed to assess the efficacy and safety of anakinra, an interleukin 1 receptor antagonist, in patients with Kawasaki disease who failed to respond to standard treatment:e.g. one infusion of 2g/kg of intravenous immunoglobulins.

DETAILED DESCRIPTION:
Kawasaki disease (KD), is the most frequent vasculitis in children before 5 years, and the main cause of acquired cardiomyopathy in adulthood. The prognosis of KD is influenced by early recognition and treatment by intravenous immunoglobulins (IVIG), which represent the standard of care and decrease significantly the risk of coronary aneurysms. Despite a first infusion of IVIG, 20% of KD patients remain febrile and are at high risk of coronary vasculitis. To date there is no agreement for a more effective second line treatment. On the basis of the autoinflammatory pattern of KD, we hypothesize that anti IL-1 blocking agents could bring a rapid and sustained effect on systemic and coronary inflammation in patients with KD.

Aim of the study

* To assess the efficacy of anakinra (IL-1R1receptor antagonist) in patients with KD who fail to respond to one infusion of IVIg (standard treatment).
* To assess the efficacy of anakinra on disease activity
* To assess the efficacy of anakinra on coronary lesions (eg: dilatation and aneurysm
* To assess the safety and tolerability of anakinra Patients and methods A Proof of concept (quasi experimental, non randomized cohort) study. This is a 3-year open-label, prospective multicenter trial of Anakinra in patients with acute KD who failed to respond to a first infusion of IVIG within 48h. Patients will be eligible to enter the study if they have persistence (or recrudescence of fever) within 48 hours after the infusion of IVIg, and if they have given their informed consent to enter the study. After appropriate screening, the study treatment will be initiated between J7 and J14 days of illness to expect full clinical effect. The only primary endpoint will be the absence of fever after 48 h of treatment (assessed at J3 of study treatment, visit 3, before the third injection of anakinra). If the patient remains febrile (fever >38°C), he will receive a double dose of anakinra (4mg/kg) at day 3 instead of 2mg/kg. Treatment will be continued until they have achieved complete response as defined in the outcome measurement section, and during a maximum of 15 days.

Expected results and expected public health benefit Anakinra treatment is expected to reduce the early and long term mortality of patients with KD, by a rapid and sustained effect on vascular inflammation. The safety of anakinra is expected to be good, as the drug has a very short half-life, which allows its rapid withdrawal in case of serious adverse event. The use of anakinra, is not associated with the risk of contamination by infectious agents, which remains even minimal, a possibility with the use of IVIG

ELIGIBILITY:
Inclusion Criteria:

* Patients, male and female, at any age ≥ 3 months (5 kg) of life, with KD according to the American Heart Association definition for complete or incomplete KD. fever ≥ 5 days and ≥ 4 of 5 main clinical signs: modification of the extremities, polymorphic exanthema, bilateral bulbar not exudative conjunctivitis, erythema of the lips or oral cavity, and cervical lymph nodes usually unilateral > 1.5 cm in diameter. In the presence of less than 4 clinical criteria and 5 days of fever, the diagnosis of disease KD is proposed in case of coronary abnormalities (at least one dilated coronary artery with internal diameter ≥ 2,5 SD from the mean normalized for body surface area (Z score) as determined by echocardiography. For indicative purpose, in case of incomplete KD, other biological supportive criteria for incomplete KD can help to ensure the diagnosis: leucocytosis, elevated CRP, elevated ESR, anaemia, hyponatremia, elevated ASAT, ALAT and gGT, hyperlipidaemia.
* Patients who failed to respond to standard therapy of KD:, e.g. Persistence or recrudescence of fever ≥ 38°C, 48 hours after the infusion of 2g/kg of IV Ig,
* Weight ≥5Kg
* Patient, parent or legal guardian's written informed consent is required
* Patient with health insurance
* Patient agrees to have effective contraception for the duration of participation in the research

Exclusion Criteria:

* Preterm and neonates, pregnancy
* Patients suspected with another diagnosis
* Patients with overt concomitant bacterial infection
* Patients previously treated with another biotherapy
* Patients with any type of immunodeficiency or cancer
* Patients with increased risk of TB infection
* Recent tuberculosis infection or with active TB

  * Close contact with a patient with TB
  * Patients recently arrived less than 3 months from a country with high prevalence of TB
  * A chest radiograph suggestive of TB
* Patients with end stage renal disease: NKF stages ≥4; eGFR≤29mL/min/1.73 m2 or diabetes mellitus or neutropenia <1500/mm3 or liver failure
* Hypersensitivity to the active substance or to any of the excipients (citric acid and anhydrous; sodium chloride disodium edetate dehydrate polysorbate 80; sodium hydroxide; water for injections)
* Patient already included in a biomedical research other than observational (e.g.; cohort, registry)

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Absence of fever | within the 48 hours after the treatment by anakinra (after the last escalation dose, if any necessary)
  The main efficacy evaluation criterion: the patient must reach a body (axillary, tympanic, oral) temperature <38 within 48 hours of treatment by anakinra (after the last escalation dose, if any necessary)

SECONDARY OUTCOMES:
Reduction in physician assessment of disease activity, on a 10 points scale, of at least to 50% | between baseline and day15
Reduction in patient's parents assessment of disease activity, on a 10 points scale, of to at least 50% | between baseline and day15
Resolution of coronary abnormalities by echocardiogram if present | at day45
CRP normalization | between baseline and day15
Adverse events frequency | between baseline and day45
  Defined with physical exam, injection tolerability, vital signs, TB risk, laboratory evaluations, echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Koné-Paut, MD, PhD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP,Bicêtre Hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Kone-Paut I, Tellier S, Belot A, Brochard K, Guitton C, Marie I, Meinzer U, Cherqaoui B, Galeotti C, Boukhedouni N, Agostini H, Arditi M, Lambert V, Piedvache C. Phase II Open Label Study of Anakinra in Intravenous Immunoglobulin-Resistant Kawasaki Disease. Arthritis Rheumatol. 2021 Jan;73(1):151-161. doi: 10.1002/art.41481. Epub 2020 Nov 17. PMID 32779863